CLINICAL TRIAL: NCT03697642
Title: A Nasopharyngeal Airway Facilitates Nasogastric Intubation in Anesthetized Intubated Patients: A Randomized Controlled Trial
Brief Title: Nasopharyngeal Airway Guide Nasogastric Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201800138A3
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-04

CONDITIONS: Nasogastric Tube; Nasopharyngeal Airway; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NG tube placement with nasopharyngeal tube (Experimental)
  Interventions: Procedure: With nasopharyngeal airway
- NG tube placement without nasopharyngeal tube (Active Comparator)
  Interventions: Procedure: Without nasopharyngeal airway

INTERVENTIONS:
Procedure: With nasopharyngeal airway — Nasopharyngeal airway is previously inserted into selected nostril. NG tube is properly lubricated and placed through Nasopharyngeal airway.
  Arms: NG tube placement with nasopharyngeal tube
Procedure: Without nasopharyngeal airway — NG tube is properly lubricated and placed into selected nostril
  Arms: NG tube placement without nasopharyngeal tube

SUMMARY:
Nasogastric tube placement is essential for various surgery and critically ill patients. However, NG tube insertion in anesthetized, paralyzed, and intubated or unconscious patients may be difficult, with reported success rate less 50% on the first attempt without any auxiliary devices. Endotracheal tube intubation narrow the space of oropharynx and hypopharynx. Loss ability to swallow and tongue drop also made the NG tube coil in the mouth easily. Investigators assume nasopharyngeal airway can facilitate NG tube insertion by opening a channel from nostril to epiglottis and reduce complications by protecting nasal cavity while inserting NG.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be > 20 years old, ASA 1~3 under going schedule general anesthesia with endotracheal tube intubation
* Patient who required NG tube placement for perioperative care

Exclusion Criteria:

* Coagulation abnormality (PLT≤100000, INR>1.2 & PT≥13)
* Hemodynamic unstable (with inotropic agent use)
* Arrythmia
* Esophageal varices or stricture, Esophageal cancer, trauma or previous esophageal surgery
* Gastric cancer involve cardiac orifice
* Corrosive chemical (strong acid or alkali) ingestion
* Skull base fracture
* Recent nasal surgery, nasal fracture or severe nasal obstruction
* Loose teeth that make endotracheal tube can not fix right side

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
First attempt successful rate | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance
Second attempt successful rate | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance
Overall successful rate insertion | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance
Time cost during NG tube placement | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance

SECONDARY OUTCOMES:
Incidence of NG tube coiling | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance during NG tube insertion
Incidence of NG tube kinking | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance during NG tube insertion
Incidence of NG tube knotting | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance during NG tube insertion
Incidence of epistaxis after NG tube placement | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance during NG tube insertion
Mean blood pressure change after NG tube placement | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance
Heart rate change after NG tube placement | can be know after NG tube placement immediately
  with or without Nasopharyngeal airway assistance

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Huang TY, Lin JR, Chung YT. A preinstalled nasopharyngeal airway in the right nasal passageway to facilitate nasogastric intubation in anesthetized and intubated patients: a prospective randomized controlled trial. BMC Gastroenterol. 2020 Nov 3;20(1):365. doi: 10.1186/s12876-020-01514-6. PMID 33143639